CLINICAL TRIAL: NCT01522495
Title: Pilot Study for: Eye vs. Spy - A Prospective, Randomized Study Evaluating Patient Outcomes With the Use of SPY Imaging During Amputations or Debridements
Brief Title: Pilot Study to Determine Percent Tissue Perfusion and Cellular Viability Using SPY Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Chief of the Division of The Center for Wound Healing, Georgetown University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Eye vs. Spy Pilot Study; 2011-114 (Other: IRB)
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SPY Imaging (Experimental): SPY Imaging Prior to Amputation or Debridements (50 participants)
  Interventions: Device: SPY Imaging, ICG dye (0.2 - 0.5 mg/kg); Device: SPY Imaging
- No SPY Imaging (No Intervention): Amputation or Debridements as Standard of Care (50 participants)
- Validation Against Angiogram (Experimental): Patients who are scheduled to undergo an angiogram will also receive ICG angiography (SPY). This will occur at specific time points: 1.) before the angiogram/intervention is performed 2.) immediately after the angiogram/intervention is performed 3.) 5-7 days after angiogram/intervention 4.) 21-30 days after angiogram/intervention.
  (30 participants)
  Interventions: Device: SPY Imaging, ICG dye (0.2 - 0.5 mg/kg); Device: SPY Imaging
- Establishing Normal Values (Experimental): To establish baseline lower extremity perfusion in non-PVD patients. Patients requiring an angiogram for other vascular processes unrelated to the lower extremity will be recruited into this study. ICG angiography (SPY) of the lower extremity will be performed at the time of the angiogram. (30 Participants)
  Interventions: Device: SPY Imaging, ICG dye (0.2 - 0.5 mg/kg); Device: SPY Imaging

INTERVENTIONS:
Device: SPY Imaging, ICG dye (0.2 - 0.5 mg/kg) — Intravenous(1X) in conjunction with SPY Imaging (1 arm)
  Other Names: Indocyanine Green, IC-GREEN
  Arms: Establishing Normal Values; SPY Imaging; Validation Against Angiogram
Device: SPY Imaging — SPY Imaging to assess tissue perfusion
  Arms: Establishing Normal Values; SPY Imaging; Validation Against Angiogram

SUMMARY:
Little is known about chronic wound microenvironments, especially in peripheral vascular disease (PVD) and diabetic patients. At the demarcation line, the percentage of viable cells and tissue is unclear. A means to determine cell viability, particularly discerning an apoptotic or necrotic cell pathway would indicate where the line of demarcation should be drawn. The information generated would better predict clinical outcome using SPY Imaging. Cellular studies are needed to successfully confirm a clear line of demarcation to eliminate surgeon subjectivity.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD), like other more central macrovascular diseases, is common in diabetes. PAD can lead to critical limb ischemia, either alone or when combined with an injury like a foot ulcer. The diabetic foot ulceration requires adequate circulation to heal; if the circulation is impaired such that the tissue oxygen demand exceeds supply, critical limb ischemia ensues, placing the limb at risk.

Most often, patients with critical limb ischemia, undergo multiple debridements in the operating room as well as vascular procedures, prior to reaching a viable level of amputation. This increases the patients' co-morbidities from repetitive exposure to anesthesia. Each debridement may be removing viable tissue and decreasing the length of the eventual amputation. Additionally, intraoperatively, the viability of the skin edges is a subjective assessment based on the surgeon's experience. That judgement can be inaccurate in 10-20% of cases and lad to reoperation. With the use of the SPY imaging system, a better assessment of not only macrovascularity, but also microvascularity of the tissues is able to be evaluated objectively. This helps identify the tissues that are underperfused.

The investigators are unaware of any literature evaluating the use of SPY imaging in the lower extremities intraoperatively during amputations or debridements. There are many studies published for the use of this technology during ophthalmic procedures , cerebral aneurismal repair, cardiac surgery and breast reconstruction. In cardiac surgery, the use of ICG based imaging has proven to be helpful in assessing the quality of bypass grafts and eliminating the need for radiography or catheter insertion (Reuthebuch et al., 2004). In ophthalmic procedures, ICG angiography has been fundamental in identifying many microvascular pathologies (Slakter, Yannuzzi, Guyer, Sorenson, & Orlock, 1995). Furthermore, neurosurgeons have found that the use of ICG angiography is far more superior than DS angiography in identifying small vessels . As it has already been proven to be a good adjunct intraoperatively to visualize microvasculature, the investigators would like to apply this to the lower extremities. Identifying underperfused tissues intraoperatively can help the surgeon objectively decide an appropriate level of amputation/debridement to effectively minimize the number of revisional surgeries. Also, there are no studies that comprehensively evaluate and compare the effectiveness of other modalities that also attempt to assess vascularity with the SPY imaging system. The information gained could be pivotal and help to gain more insight in patients with difficult to heal wounds, especially in the presence of PVD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years or older.
* Subject has PVD demonstrated by angiogram.
* Subject is undergoing the first amputation/debridement after vascular intervention, if intervention is/was warranted.
* Subject has had a vascular consult and/or intervention.
* Subject must sign an IRB approved informed consent.
* Subject is willing and able to complete required follow up.

Exclusion Criteria:

* Subject has no evidence of PVD
* Subject's wound presents with a malignancy in the wound bed.
* Subject has liver disease (Previously diagnosed with liver disease or elevated AST, ALT, Alk Phos, or Bilirubin labs within 30 days of procedure).
* Subject has a disorder or situation that the investigator believes will interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Determination of percent cellular viability | 6 weeks
  Determine percent cellular viability (vs. apoptotic/dead) of cells at demarcation line
Rate of infection, dehiscence and re-amputation | 20 weeks
  Rate of infection, dehiscence and re-amputation in patients undergoing SPY imaging
Number of debridements, revisional surgeries and days of stay in hospital | 20 weeks
  The endpoint for evaluation will be the number of revisional surgeries and number of days of stay in hospital within 20 weeks of the first procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Attinger, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center; Center for Wound Healing, Washington D.C., District of Columbia, United States